CLINICAL TRIAL: NCT00500435
Title: A Pilot Study of Laparoscopic Extraperitoneal Lymph Node Dissection in Patients With Locally Advanced Cervical Cancer
Brief Title: Extraperitoneal Lymph Node Dissection in Patients With Cervical Cancer
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: ID03-0098
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer; Laparoscopy; Lymph Node Dissection; Extraperitoneal Laparoscopic Lymphadenectomy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Laparoscopy Procedure: Laparoscopy procedure in abdomen to remove para aortic lymph nodes of patients diagnosed with cervical cancer.
  Interventions: Procedure: Extraperitoneal Laparoscopic Lymphadenectomy

INTERVENTIONS:
Procedure: Extraperitoneal Laparoscopic Lymphadenectomy — Laparoscope used to find and remove para aortic lymph nodes in abdomen.

SUMMARY:
Primary Objectives:

* To determine the feasibility of performing an extraperitoneal laparoscopic lymphadenectomy in patients with stage IB2-IVA cervical carcinoma who are dispositioned to undergo radiotherapy and concurrent chemotherapy.
* To document intraoperative and postoperative complications in patients undergoing extraperitoneal laparoscopic lymphadenectomy.
* To determine the rate of lymph node metastases in the para-aortic region in patients with stage IB2-IVA cervical cancer.
* To correlate histopathological findings in the para-aortic lymph nodes with preoperative imaging studies (Positron emission tomography (PET) and magnetic resonance imaging (MRI) and computed tomography (CT)).

DETAILED DESCRIPTION:
Currently, the decision about how much radiation should be given to patients with stage IB2-IVA cervical cancer is based on direct physical examination, chest x-ray, computed tomography (CT) scan, magnetic resonance imaging (MRI) scan, cystoscopy (examination of the bladder), proctoscopy (examination of the rectum), and possibly an intravenous pyelogram (a test that uses dye to outline the bladder, kidneys, and the tubes that carry urine from the kidney to the bladder on an x-ray). Unfortunately, these techniques may not identify cancer that has spread to the lymph nodes. Studies have shown that cancer in the lymph nodes is one of the most important factors in the return of the cancer. Standard radiation therapy treats the lymph nodes in the pelvis area but does not include the lymph nodes in the abdomen (called para aortic lymph nodes) . If cancer is present in the lymph nodes in the abdomen and it was not detected by the standard techniques, the cancer could be undertreated and the risk of the cancer returning would be high.

Using a surgical procedure called extraperitoneal laparoscopic lymphadenectomy, surgeons can remove and examine the lymph nodes in the abdomen. This may help to find cancer in the lymph nodes that cannot be detected using standard techniques. If these lymph nodes contain cancer, the area of the body treated with radiation can be "extended" to treat new areas. This means that radiation will be used to treat both the para-aortic lymph nodes (lymph nodes in the abdomen) in addition to the standard pelvic radiation.

Before beginning your radiation therapy, you will be taken to the operating room for the laparoscopy procedure. The laparoscopy procedure involves placing a telescope-like instrument through a small, usually ½ inch, incision (cut) in the abdomen. Three other small incisions are made to place additional instruments that may be needed to complete the surgery. Before the laparoscope is inserted, carbon dioxide gas (CO2) is introduced into the side of the abdomen. This gas helps to separate the organs inside the abdominal cavity, making it easier for the surgeon to see. The laparoscope is then inserted through the small incision. The laparoscope has a small camera on the end of the instrument. This is attached to a high-resolution TV monitor. Using the TV monitor, the surgeon can see inside your body without making a large incision. While watching the TV monitor, the surgeon uses the laparoscope to find the para aortic lymph nodes and removes them. Once the procedure is finished, the carbon dioxide gas is removed and you are taken to the recovery room.

The lymph nodes that were removed will be sent to the lab and evaluated for the presence of any cancer cells. If cancer is found, your radiation therapy will be adjusted to also treat the lymph nodes. If no signs of cancer is found, you will receive the standard radiation therapy.

If, during the laparoscopy procedure, the surgeon finds an obvious sign of cancer (such as enlarged lymph nodes) then an exploratory laparotomy will be performed. This procedure involves making a long incision in the abdomen so that the surgeon can remove any additional lymph nodes that may contain cancer.

All participants will undergo a Positron Emission Tomography scan, also called a PET scan, before their scheduled surgery. This test studies the function of organs such as the heart, brain, and bone. The test is different from other imaging tests such as x-rays, CT scans, or MRI's because PET images show how tissues function. The other imaging methods show what the tissues look like. The PET scanner is similar to a CT or an MRI scanner. The bed on the scanner moves during the exam so that each area of the body can be imaged. The PET scanner makes no noise.

Before the PET scan, a blood test (about 1 teaspoon) will be done to check your blood sugar level. The day before the scan, you will be asked to follow a special diet. This is to control the amount of sugar in your bloodstream. One the day of the scan a small tube will be placed in your vein to administer a very small amount of radioactive material. This material allows the PET scanner to "see" where the sugar is metabolized in your body. The amount of time the scan takes depends on how tall you are and why you are having the test. After the scan, patients rest for about 45 to 90 minutes before being discharged. Family members are not allowed to come in with the patient during the test. Overall, you should allow about 3 hours for this scan. If you had this test prior to entering the study, you do not have to have this test repeated as long as it was done within 4 weeks of the laparoscopy.

This is an investigational study. The PET/CT scan will be performed only at M. D. Anderson and the laparoscopy procedure will be performed at both M. D. Anderson and Lyndon Baines Johnson General Hospital (LBJGH). The chemotherapy and/or radiation treatments may be done at either MD Anderson or in your hometown. Up to 70 patients will be enrolled in this multicenter study. Up to 55 will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage IB2-IVA cervical cancer who are candidates for treatment with radiotherapy and concurrent chemotherapy.
* Patients with biopsy-proven cervical carcinoma, any histology.
* Patients must have no evidence of para aortic lymphadenopathy (< 2cm in diameter) on the preoperative computed tomography (CT) or magnetic resonance imaging (MRI) scan of the abdomen and pelvis.
* Patients must sign an IRB approved informed consent.
* Patients with adequate bone marrow, renal and hepatic function: White Blood Count (WBC) >/= 3,000 cells/mcl, Platelets >/= 100,000/mcl, Creatinine </= 2.0 mg%, Bilirubin </= 1.5 x the upper limit of normal and Serum glutamic pyruvic transaminase (SGPT) </= 3 x the upper limit of normal.
* Zubrod Performance Status of 0, 1, or 2.
* Patients must be suitable candidates for surgery.
* Patients who had a PET/CT scan prior to study entry are eligible if a) the study was done within 4 weeks of surgery, and b) they have no evidence of para aortic lymphadenopathy (< 2cm in diameter) on either a preoperative CT or MRI scan of the abdomen and pelvis.

Exclusion Criteria:

* Patients who have had prior retroperitoneal surgery.
* Patients who have received prior pelvic or abdominal radiotherapy.
* Patients known to have upper abdominal intraperitoneal disease or evidence of ovarian metastases.
* Patients who are pregnant.
* Patients with evidence of distant metastases on chest x-ray, CT or MRI scan or by physical examination.
* Patients with contraindications to laparoscopy.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with stage IB2-IVA cervical cancer.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2003-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Complication Rates | 6 Years
  Complication rates determined as number of participants with inherent complications to procedure calculated separately from overall complications divided by to total number of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Ramirez, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - UT MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org